CLINICAL TRIAL: NCT02560662
Title: PhysSurg-B : Physical Activity in Relation to Surgical Operations, a Prospective Open-label Randomized Controlled Multicenter Study of the Effect of Physical Activity on Recovery After Breast Cancer Surgery
Brief Title: PhysSurg-B : Physical Activity in Relation to Surgical Operations - Breast Cancer
Acronym: PhysSurg-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Roger Olofsson Bagge, MD, PhD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PhysSurg-B
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer, physical exercise, recovery
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity (Experimental): Individual consultation with a physiotherapist in order to increase the participants existing level of physical activity by adding 30minutes of physical activity daily, preoperatively and 4 weeks postoperatively.
  Interventions: Behavioral: Physical activity
- Control (No Intervention): Participants randomized to the control group will not be advised to change their current level of physical activity.

INTERVENTIONS:
Behavioral: Physical activity — Preoperative intervention - takes place from randomization until surgery (4 weeks +/-2 w):
  • 30 minutes of exercise daily added to the existing daily exercise routine. The level of exercise should produce shortness of breath but the patient should be able to talk without much effort.
  Postoperative intervention - takes place from discharge from the hospital until 4 weeks postoperatively:
  • 30 minutes of exercise daily added to the existing daily exercise routine. The level of exercise should produce shortness of breath but the patient should be able to talk without much effort.
  Participants randomized to intervention will receive a visit to a physiotherapist for personally adjusted information regarding the intervention, later followed up with a telephone call.
  Arms: Physical activity

SUMMARY:
The purpose of this study is to investigate whether a training program with intensified physical exercise prior to and after surgery for breast cancer enhances postoperative recovery.

DETAILED DESCRIPTION:
This study is designed as a randomised, controlled, non-blinded multicenter trial with two parallell study groups, intervention and control. The primary endpoint of recovery is measured within 12 months after surgery.

After randomisation, participants in the intervention group will be scheduled for an individual consultation with the physiotherapist, where the are advised to increase their Daily physical activiy level with an additional 30 minutes. The added physical activity is registered in an exercise diary daily.

All included participants will be asked to complete questionnaires at inclusion (I), 4 weeks (+/- 1 w) postoperatively (II) and 12 months (+/-1 month) postoperatively (III).

Data regarding patient characteristics, surgical details, postoperative events, complications according to Clavien - Dindo and additional treatment will be collected using eCRF: (I) 30 Days postoperatively, (II) 90 days postoperatively and (III) 12 months postoperatively. Data will also be retrieved from the Swedish National Breast Cancer Register, the Swedish Social Insurance Agency and the Swedish National Death Register.

Patrticipants who wish to be excluded from the study will be asked if already collected data may be analysed in the study.

The code for the study cohort will include personal identity as well as a study specific code. This is placed on a server, with limited access, at Sahlgrenska University Hospital. The database is placed on a server within the University of Gothenburg system accessible with username and code. The database includes only the study specific code for each participant. Data from questionnaires will be entered manually. Length of hospital stay will be acquired from the hospital registries and then entered manually into the database. Data from CRF (I-III) will be entered in the same database, as well as data retrieved from the Swedish National Breast Cancer Register, the National Death Register and Swedish Social Insurance Agency.

In all a high security standard with automatic back up of server data is present as well as firewalls against external violation. A data manager, employed by the SSORG unit will be responsible for the database.

The investigators plan to perform an interim analysis for the first 100 patients included, in order to make a more exact estimate of the power needed. An external monitoring committee will be appointed for the interim analysis, and the question to the committee will be limited to a recalculation of cohort size.The participants will be analysed according to randomisation (intention to treat-type of analysis).

ELIGIBILITY:
Inclusion Criteria:

* All female patients at the participating hospital scheduled for breast cancer surgery will be asked to participate.

Exclusion Criteria:

* Inability to understand given information.
* Inability to perform the intervention, as assessed by the person performing inclusion.
* Withdrawal of informed consent.
* Male sex.
* Stage IV breast cancer at diagnosis.
* Neoadjuvant breast cancer treatment.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Change in self-reported physical and psychological recovery | Inclusion, 4 weeks (+/- 1 week) and 12 months (+/- 1 month) postoperatively
  Measured using validated questions within a questionnaire
Sick leave | 12 months postoperatively
  Data from the Swedish Social Insurance Agency (Försäkringskassan) on total number of days and the reasons (diagnosis) for any sick-leave episodes

SECONDARY OUTCOMES:
Length of hospital stay | 30 days postoperatively
  For each participant the number of days of hospital stay for the index surgery will be collected
Adverse events | 90 days postoperatively
  Classified according to Clavien-Dindo
Re-operations and re-admittances | 12 months postoperatively
  The number of participants with re-admittances to hospital and/or re-operations after the index surgery will be retrieved from hospital registration systems and analyzed
Mortality | 3 and 5 years postoperatively
  Data retrieved from National Death Register, overall and cancer-specific mortality
Health economy | 12 months postoperatively
  Analysis using modelling, focusing on the societal perspective and measuring the effects of regular physical exercise for resource consumption, measured in Swedish currency SEK.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Olofsson Bagge, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heiman J, Onerup A, Bock D, Haglind E, Olofsson Bagge R. The effect of nonsupervised physical activity before and after breast cancer surgery on quality of life: Results from a randomized controlled trial (PhysSURG-B). Scand J Surg. 2022 Dec;111(4):75-82. doi: 10.1177/14574969221123389. Epub 2022 Sep 15. PMID 36113110
- [Derived] Heiman J, Onerup A, Wessman C, Haglind E, Olofsson Bagge R. Recovery after breast cancer surgery following recommended pre and postoperative physical activity: (PhysSURG-B) randomized clinical trial. Br J Surg. 2021 Jan 27;108(1):32-39. doi: 10.1093/bjs/znaa007. PMID 33640941